CLINICAL TRIAL: NCT02253004
Title: The Effect of the Selective PDE3 Inhibitor on Migraine With Aura Induction and Vascular Endothelial Function.
Brief Title: Induction of Migraine Aura With Cilostazol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Christina Kruuse, Associate professor, consultant neurologist, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-3-2013-166; 2013-004188-29 (EudraCT Number)
Record Dates: First submitted 2014-09-26; First posted 2014-10-01 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Migraine With Aura; Stroke
MeSH Terms: conditions — Migraine with Aura; Stroke | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Cilostazol 200 mg single dose
  Interventions: Drug: Cilostazol
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol — Single oral administration of active or placebo one week apart
  Other Names: Pletal
  Arms: Active
Drug: Placebo
  Arms: Placebo

SUMMARY:
In a double blind placebo-controlled cross-over study the effect of cilostazol on aura induction and endothelial response is tested in patient with migraine with aura.

DETAILED DESCRIPTION:
Migraine with aura is associated to an increased risk of stroke. The mechanism behind such increased risk is not fully understood. Cilostazol induce headache and migraine in migraine patients and is used as secondary prevention of stroke. The effect on aura induction is not known. We investigate the aura inducing potential of cilostazol and associated changes in endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with aura
* Minimum of 2 attacks/year

Exclusion Criteria:

* Chronic tension type headache
* Cardiac arrhythmias

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Aura | 24 hours
  Induction of aura reported by an aura diary for 24 hours post medication

SECONDARY OUTCOMES:
Migraine | 24 hours
  Induction of headache resembling usual migraine attacks
Endothelial response | 3 hours
  Measurement of endothelial response by Endopat2000 before and after administration of placebo and cilostazol

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kruuse, MD PhD DMSc, Principal Investigator — Consultant Neurologist, Dept Neurology
Locations (1):
- Herlev Hospital, Dept Neurology, Herlev, Denmark